CLINICAL TRIAL: NCT04777578
Title: Effects of Dry Needling in Teres Major in Patients With Shoulder Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Luis Ceballos Laita, Clinical professor, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CASVE-NM-21-504
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DN (Experimental)
  Interventions: Other: Dry needling
- Control (No Intervention)

INTERVENTIONS:
Other: Dry needling — Dry needling based on fast-in fast-out technique in the teresa major muscle
  Arms: DN

SUMMARY:
The aim of the study is to investigate the effects of the dry needling technique in teres major muscles on pain, range of motion, strength and extensibility of the posterior part of the tissues of the shoulder in athletes with shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* Athletes with Shoulder pain
* Glenohumeral internal rotation deficit
* Presence of active MTrP in the teres major muscle

Exclusion Criteria:

* Previous surgery in the upper limb
* Previous physiotherapy treatments in the shoulder
* Dry needling contraindications
* Previous dry needling experience to mantain the blinding

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-12-20 (Estimated); Study Completion 2022-01-05 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Baseline
  the examiners assess the pain intensity using a visual analoigue scale
Pain intensity | immediately after the intervention
  the examiners assess the pain intensity using a visual analoigue scale

SECONDARY OUTCOMES:
Range of motion | Baseline
  the examiners assess the shoulder range of motion with an universal goniometer
Range of motion | immediately after the intervention
  the examiners assess the shoulder range of motion with an universal goniometer
Strength | Baseline
  the examiners assess the shoulder range of motion with a hand-held dynamometer
Strength | immediately after the intervention
  the examiners assess the shoulder range of motion with a hand-held dynamometer
Extensibility | Baseline
  the examiners assess the extensibility of the posterior part of the tissues of the shoulder using a digital inclinometer
Extensibility | immediately after the intervention
  the examiners assess the extensibility of the posterior part of the tissues of the shoulder using a digital inclinometer

CONTACTS AND LOCATIONS:
Locations (1):
- Luis Ceballos Laita, Soria, Spain

IPD SHARING:
Plan to Share IPD: Undecided